CLINICAL TRIAL: NCT05722834
Title: Self-regulation for Older Adults With Asthma Through Remote Education
Acronym: SOAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Principal Investigator, Alan Baptist, Associate Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00219528
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: Asthma education; Self-Regulation; Remote education; Counseling
MeSH Terms: conditions — Asthma; Self-Control

STUDY DESIGN:
Intervention Model Description: 12 participants along with the Primary care physicians will be enrolled (both will sign consents).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SOAR intervention (Experimental): The SOAR intervention will be a remote intervention that will follow a self-regulation process in which the participant first selects a specific problem to address and researches how asthma is preventing resolution of the problem, and finally identifies and develops a plan to achieve the objective.
  Interventions: Behavioral: SOAR intervention

INTERVENTIONS:
Behavioral: SOAR intervention — This program intervention will be over 6 weeks and participants will have two group sessions and individual sessions, all conducted by an asthma health coach over Zoom (or phone). The two Zoom group sessions will be recorded so that all the information from the conversations will be maintained and used for research purposes. Additionally, participants will keep track of asthma symptoms and complete surveys at specified time-points (the last one at 6 months after participation).
  Primary care physicians will be sent emails regarding the self-management goals of their patients.

SUMMARY:
This research is studying whether changing an individual's behaviors may have an impact as a treatment or outcome for asthma.

The purpose of this study is to implement and evaluate an asthma self-management intervention through multiple locations in the United States that is tailored to the challenges older adults face and is based on an individual behavioral theory of change.

Eligible participants will be enrolled and participate for six weeks in the SOAR intervention.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma
* Poorly controlled asthma, as evidenced by a score ≤ 19 on the Asthma Control Test
* Have a primary care provider willing to participate in the study by receiving email updates regarding the status of the participant

Exclusion Criteria:

* Physician diagnosis of any other significant cardiopulmonary disease (including chronic obstructive pulmonary disease)
* A greater than 20 pack-year smoking history
* Lack of telephone access
* Decreased cognitive capacity such that participation in the program would not be possible

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The Feasibility of Intervention Measure (FIM) of the SOAR intervention for patients and providers | Day 43
  A 4-item instrument to assess perceived intervention feasibility. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean. Higher scores indicate greater perceived feasibility.
Acceptability of Intervention Measure (AIM) of the SOAR intervention for patients and providers | Day 43
  A 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean. Higher scores indicate greater perceived acceptability.
Intervention Appropriateness Measure (IAM) for patients and providers | Day 43
  This is a 4-item measure of perceived intervention appropriateness. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean. Higher scores indicate greater perceived appropriateness.

SECONDARY OUTCOMES:
Change in Asthma control will be determined with the Asthma Control Test (ACT) | baseline to 6 months
  Asthma Control Test (ACT) has 5 questions. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Change in Perceived Control of Asthma Questionnaire (PCAQ) | baseline to 6 months
  This questionnaire has 11 questions. Responses are graded on a 5-point scale, scoring between 11 and 55, with higher scores reflecting greater perceived control of asthma.
Change in Health Care Communication Questionnaire (HCCQ) | baseline to 6 months
  This is a 6-question questionnaire. Responses are given on a Likert scale from Strongly Disagree to Strongly Agree. The range of scores is 1-7, the final score being the mean of all individual responses. Higher scores indicate a perception of better communication with the health care provider.
Change in Geriatric Depression Scale - Short Form (GDS-SF-15) | baseline to 6 months
  This is a 15-question instrument that has a range from 0-15. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Change in Mini Asthma Quality of Life Questionnaire (AQOL) | baseline to 6 months
  This is a 15 question questionnaire. The scores range 1-7, with higher scores indicating better quality of life.
Change in Short Form Health Survey (SF-12v2) - 12 questions. Survey responses are grouped into two scales: physical score and mental score. Higher scores indicate perception of better health. | baseline to 6 months
  This is a 12 question survey. Survey responses are grouped into two scales: physical score and mental score. The range of scores is 0-100, higher scores indicate perception of better health.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Baptist, MD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Illinois-Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No